CLINICAL TRIAL: NCT05047276
Title: Phase I/II Study of AloCelyvir in Patients With Metastatic Uveal Melanoma
Acronym: PULSE-UM
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: José María Piulats Rodríguez (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, José María Piulats Rodríguez, Sponsor's representative, Institut d'Investigació Biomèdica de Bellvitge
Organization: Institut d'Investigació Biomèdica de Bellvitge (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PULSE-UM
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Uveal Melanoma, Metastatic
Keywords: Uveal Melanoma, Advanced therapy, AloCelyvir, Icovir-5, Mesenchymal Stem Cells, Oncolytic virus
MeSH Terms: conditions — Uveal Melanoma; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AloCelyvir (Experimental): Delivery of Icovir-5 by mesenchymal carrier cells in uveal melanoma patients with hepatic metastases.
  Interventions: Biological: AloCelyvir

INTERVENTIONS:
Biological: AloCelyvir — Delivery of Icovir-5 by mesenchymal carrier cells in uveal melanoma patients with hepatic metastases.

SUMMARY:
This is a non-randomized, single arm, single center, phase I/II study of AloCelyvir in subjects with mUM to the liver, the main site for M1 in this disease. This study is divided into 3 phases: Screening, Treatment, and Follow-up. After informed consent is obtained, subjects will enter in the Screening phase to assess eligibility criteria and perform a mandatory tumor biopsy. Upon meeting criteria, eligible subjects will be entered into the Treatment phase. Patients will receive AloCelyvir in weekly intravenous infusions at doses of 0.5x106 cells/kg for 8 weeks. After 4 first treatment doses a new tumor biopsy will be mandatory. Treatment will be maintained for 2 months (8 weeks) but can be stopped earlier if disease progression, unacceptable toxicity, or patient withdrawal. Subjects that are no longer receiving AloCelyvir will enter the Follow-up phase. Subjects that are no longer receiving AloCelyvir because of unacceptable toxicity or due to investigator judgment will undergo radiological evaluations of the tumor every 8 weeks during the first 12 months (48 weeks), and then every 12 weeks until the progression of disease (progression follow-up). Subjects that are no longer receiving Alocelyvir because of progression will enter the long term OS follow-up until their death or until the end of the study, whatever happens before. Subjects who have switched to an alternative treatment without disease progression will receive a formal follow-up with images tests until progression, and after progression long term follow up to record the date of death.

DETAILED DESCRIPTION:
0. Background:

Uveal melanoma (UM) is an orphan neoplasm but it is the most common primary intraocular malignant tumor in adults. Global overall survival (OS) at 5 years is lower than 50%. This elevated mortality rate is caused by a high incidence of metastases, and lack of active therapy. The metastatic behavior differs from cutaneous melanoma (CM) given the purely hematogenous dissemination and the tendency to metastasize to the liver 3. When liver metastases develop, life expectancy is reduced to 8-9 months. Chemotherapy treatment is unsuccessful in metastatic UM (mUM) and results in less than 5% overall response rate (ORR). There is no proof that chemotherapy prolongs survival and the 5-year survival rate of patients with UM has not improved in 25 years . New targeted therapies have not improved results.

The PULSE-UM study plans to treat mUM patients with an advanced therapy that seeks to activate the immune system and to study the mUM immune-environment in different ways to identify new immunotherapy targets.

1. Overview of study design.

   This is a single arm, single center, phase I/II study of AloCelyvir in subjects with metastatic uveal melanoma with liver disease. This study is divided into 3 phases: Screening, Treatment, and Follow-up. After informed consent is obtained, subjects will enter the Screening phase to assess eligibility criteria and perform a mandatory tumor biopsy. Upon meeting criteria, eligible subjects will be entered into the Treatment phase. Patients will receive a weekly infusion of AloCelyvir. New tumor biopsy will be mandatory and performed around day +28 +/- 3 days (week 4). Treatment will be administered for 8 consecutive weeks but can be stopped because disease progression, unacceptable toxicity or patient withdrawal. Subjects that have finished the 8-weeks period or has stopped the treatment because of unacceptable toxicity or due to investigator judgment will enter the follow-up phase (firstly for PFS until progression and lately long term follow-up until death).

   Subjects that have finished the 8-weeks period or has stopped the treatment because of unacceptable toxicity or due to investigator judgment will undergo radiological evaluations of the tumor every 8 weeks during the first 12 months (48 weeks), and then every 12 weeks until the progression of disease (progression follow-up). Also, patients that have received at least 1 dose of AloCelyvir will also initiate the safety evaluations. Safety evaluations will performed be every 8 weeks during the first 12 months (48 weeks).

   Subjects that are no longer receiving AloCelyvir because of progression will enter the long term OS follow-up until their death or until the end of the study (whatever happens before).

   Subjects who have switched to an alternative treatment without disease progression will receive a formal follow-up with images tests until progression, and after progression long term follow up to record the date of death.
2. Screening phase.

   Screening will occur between Day -28 and Day 0 that is before first treatment administration. The purpose of the screening period is to establish protocol eligibility, as specified in the inclusion/exclusion criteria.

   Informed consent of study procedures and tumor biopsy sample should be obtained prior to the 28-day screening window after the study has been fully explained to each subject, in order to permit tumor biopsy sample acquisition and analysis prior to enrollment.

   If laboratory or imaging procedures were performed for alternate reasons prior to signing consent, these can be used for screening purposes with consent of the patient. However, all screening laboratory and imaging results must have been obtained within 28 days of enrollment.

   A mandatory fresh tumor tissue from liver biopsies before starting therapy, to compare stromal cell populations after combination treatment with AloCelyvir should be collected during screening visit (after informed consent is signed by the patient) and managed according to what is detailed in the laboratory manual. The collection of baseline tumor biopsies and around day +28 (week 4) is mandated unless the procedure confers a risk to the patient. The collection of tumor biopsies at the time of progression is optional but strongly encouraged.

   Results of screening assessments must be obtained prior to the first dose of study drug (Cycle 1/Day 1). Assessments may be performed on Day -1 or on Cycle 1/Day 1 prior to dosing. Clinical laboratory tests including pregnancy test (where applicable) can be performed within 72 hours prior to the first dose of study drug. Subjects who complete the baseline visit and continue meeting the inclusion/exclusion criteria will begin the treatment phase of this study.
3. Treatment phase.

   The treatment phase will begin at the time of enrolment of the first patient and will consist in 2 cycles of 4 weeks (28 days). The treatment phase will end when the last patient finishes treatment plant.

   Once registered and having received the confirmation of enrolment form from eCRF, subjects will receive a weekly IV infusion of AloCelyvir 0.5x106 cells/kg.

   Treatment will continue for 8 weeks or until confirmed disease progression, unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met. Any grade 3 or grade 4 toxicity according to CTCAE criteria will be discussed in a safety committee formed by Principal Investigator, the head of UICEC Pharmacovigilance Team and the Clinical Trial Unit at IDIBELL. This committee will deem the toxicity as unacceptable or not.

   Every effort should be made to minimize the time between enrollment and starting treatment. (i.e. within 2 day of enrollment).

   An additional mandatory fresh tumor tissue from liver biopsies on day +28 +/- 3 days should be collected to compare stromal cell populations after combination treatment AloCelyvir. Management of sample is detailed in the laboratory manual.

   Results for LFTs, full blood count, and creatinine must be available before commencing an infusion of AloCelyvir, and reviewed by the treating physician or Investigator prior to dosing/dispensing.

   Subjects will be visited by Investigators every other week during the treatment phase, to closely follow up toxicity. Patients should be visited at least every month thereafter and every time that Principal Investigator deemed necessary.

   Subjects will undergo radiological evaluations of the tumor every 8 weeks during the first 48 weeks and then, every 12 weeks until disease progression. This schedule MUST be followed regardless of any delays in dosing or end of treatment due to other reason than disease progression.

   Safety assessments will be performed at each visit and include patient interview and reviewing of additional source documentation such as investigations, medical history and concomitant medications, as needed.
4. End of treatment visit.

   The visit scheduled 4 weeks after AloCelyvir last planned dose will be considered the end-oftreatment visit. This visit should be scheduled for 28 +/-3 days after the end of treatment for any reason.
5. Progression (PFS) follow up.

   Patients that end treatment due to any reason other than disease progression, according to RECIST 1.1, will follow tumor evaluations every 8 weeks (up to week 48) and every 12 weeks or clinically indicated thereafter, until disease progression.
6. Long term follow-up phase.

   All patients (both, after disease progression or in the case that patients have switched to an alternative treatment without documented progression), should be followed until death or study closure. Date and reason of death should be documented consistently in patient record and in the eCRF.
7. Study oversight for safety evaluation.

This protocol will contain a safety part followed by an expansion part. The first 3 patients will be included in the safety part. Due to lack of standard treatment and dismal prognostic in this disease, no time restriction between patient enrollment will be applied.

When all these 3 patients received at least 4 AloCelyvir administrations, the Principal Investigator together with the head of the Pharmacovigilance Team of the UICEC and the Clinical Trial Unit at IDIBELL will discuss and review the reported toxicity. If no grade 3 or grade 4 toxicity was presented, the safety part will be closed and then the expansion part will begin. If a grade 3 toxicity was presented and after the team evaluation, another 3 patients will be included in the safety part. The same toxicity evaluation will be applied in this new safety part.

Patients in both the safety and the expansion part will have a weekly visit during treatment phase followed by the end-of-treatment visit. Onwards, all patient will enter in the progression follow-up phase. In this phase, along with the progression visits, patients will also have the safety evaluation. Safety evaluations will be performed every 8 weeks (after the las dose of AloCelyvir) during the first 48 weeks.

A subject may elect to discontinue AloCelyvir at any time for safety, medical, or personal reasons. Patients who choose to discontinue study drug prior to the end of the 8-weeks treatment period will be followed in the progression follow up period and continue to undergo regularly scheduled disease assessment until documentation of disease progression or start of an alternative anticancer treatment. Also, patients that have received at least 1 dose of AloCelyvir will also initiate the safety evaluations.

All subjects will be followed for overall survival and all post progression cancer treatments administered will be recorded. Subjects may at any time, withdraw consent for further study participation. A subject who has ceased to return for visits will be followed up by mail, phone, or other means as much as possible to gather information such as the reason for failure to return and the status of treatment compliance, presence or absence of adverse events, and clinical courses of signs and symptoms, and the information will be recorded in the eCRF.

Subjects who early withdrew from the study or treatment will be discontinued for 1 of these primary reasons: adverse event(s), lost to follow-up, subject choice, progressive disease, or administrative/other. In addition to the primary reason, the subject may have indicated 1 or more of these reasons as secondary reasons for discontinuation. Study disposition information will be collected on the appropriate eCRF. A subject removed from the study for any reason may not be replaced.

Safety will be assessed by monitoring and recording all AEs including all CTCAE grades (for both increasing and decreasing severity) and serious adverse events (SAEs); regular monitoring of hematology and clinical chemistry; physical examinations; and regular measurement of vital signs, and electrocardiograms (ECGs) as detailed in the schedule of visits and procedures.

Safety evaluation will be performed by PI in each visit, all findings will be collected in the eCRF and, when applicable, will be expedited informed to Sponsor according to what is detailed in Assessment of Safety section. Coordinating Investigator will be the principal contact in IDIBELL for pharmacovigilance surveillance and will be informed by the UICEC of each new SAE received and will participate on the management of study emergent toxicities. Furthermore, a monthly report with all new SAE reported by sites will be distributed both, to sites and Sponsor. Annual Safety Reports (DSUR) will be elaborated with the cumulative safety information of the trial and submitted to Coordinating Investigator, Sponsor and Industry Partner, before sending to Competent Authorities as required by current regulation for clinical trials.

Additionally, the Principal Investigator together with the head of the Pharmacovigilance Team of the UICEC and the Clinical Trial Unit at IDIBELL will meet monthly to discuss all SAEs reported . They will meet also every time a Grade 3-4-5 toxicity is reported to asses causality to AloCelyvir and oversight safety profile of the Study. Also, the will meet after the 3 first patients in the safety part of the study have received the first 4 infusions of AloCelyvir.

If at any time safety profile of the study is not acceptable, corrective measures will be implemented by the Sponsor, otherwise the study would be halted.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed metastatic uveal melanoma with measurable disease not eligible for curative therapy.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for nonnodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, PET/CT, MRI, or calipers by clinical exam. Patients must have at least 1 biopsiable liver metastasis.
* Patients can have received prior therapy for metastatic disease, excepting for treatments listed in exclusion criteria.
* Patients must be 18 years of age or older at time of study entry.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations not performed according to normal practice. Patient must consent for liver metastasis biopsies donation at day 0 and day +28 since treatment initiation.
* Adequate normal organ and marrow function as defined below:

  * Haemoglobin ≥9.0 g/dL
  * Absolute neutrophil count (ANC) > 1.5 x 109/L (> 1500 per mm3)
  * Platelet count ≥ 100 x 109/L (>100,000 per mm3)
  * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with Coordinating Investigator.
  * Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤3 x ULN.
  * Creatinine clearance ≤1.5 x ULN or a calculated by Cockcroft-Gault >60 ml/min/1,73.
* Female participant has a negative serum pregnancy test prior to revieving study treatment if of childbearing potential and agrees to abstain from activities that could result in pregnancy from screening through 150 days after the last dose of study treatment, or is of non-childbearing potential.
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential as confirmed by a negative urine or serum pregnancy test within 7 days prior to inclusion. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Amenorrheic for ≥1 year in the absence of chemotherapy and/or hormonal treatments,
  * Luteinizing hormone (LH) and/or follicle stimulating hormone and/or estradiol levels in the post-menopausal range,
  * Radiation induced oophorectomy with last menses >1 year ago,
  * Chemotherapy induced menopause with >1 year interval since last menses,
  * Surgical sterilization (bilateral oophorectomy or hysterectomy).
* Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
* Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Male participants are eligible to participate if they agree to the following during the intervention period and for at least 120 days after the last dose of study intervention:

  * Refrain from donating sperm, PLUS either:
  * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent, OR
  * Must agree to use contraception, unless confirmed to be azoospermic (vasectomized or secondary to medical cause ), as detailed below:
  * Agree to use a male condom plus partner use of an additional contraceptive method when having penile-vaginal intercourse with a WOCBP who is not currently pregnant. Note: Men with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or use a male condom during each episode of penile-vaginal penetration.
  * Male participants must agree to use male condom when engaging in any activity that allows for passage of ejaculate to another person of any sex.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Must have a life expectancy of at least 12 weeks.

Exclusion Criteria:

* Prior treatment with Celyvir or AloCelyvir. Previous treatment with immune checkpoint blockaders (E.g. anti-PD1/PDL1 or anti CTLA4) are permitted.
* Prior malignancy except for any of the following:

  * Carcinoma in situ or non melanoma skin cancer.
  * Any prior malignancies ≥3 years before randomization with no subsequent evidence of recurrence or progression regardless of the stage.
  * Stage 0 or Stage 1 cancer <3 years before randomization that has a remote probability of recurrence or progression in the opinion of the investigator.
* Patients with brain or leptomeningeal involvement should be clinically stable with unchanged or descendant steroids (≤10mg/day of prednisone or its equivalent) for at least 2 weeks.
* Patients weighing <30kg will be excluded from enrollment.
* Participation in another clinical study with an investigational product during the last 4 weeks.
* Concurrent enrolment in another clinical study, unless it is an observational (noninterventional) clinical study or during the follow-up period of an interventional study.
* Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) ≤28 days prior to the first dose of study drug If sufficient wash-out time has not occurred due to the schedule or PK properties of an agent, a longer wash-out period will be required, as agreed by Sponsor designated Coordinating Investigator and Principal Investigator.
* Any unresolved acute toxicity NCI CTCAE Grade ≥3 from previous anticancer therapy.
* Any concurrent chemotherapy, IMP, biologic, or hormonal therapy for cancer treatment different to AloCelyvir. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
* Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
* Major surgery within a minimum of 2 weeks prior to inclusion; patients must have recovered from any effects of any major surgery prior to inclusion. Note: Local surgery of isolated lesions for palliative intent and minor surgeries performed to obtain biological material for the study (i.e. liver biopsy) are acceptable.
* History of allogeneic organ transplantation.
* Active and prior serious documented autoimmune or inflammatory disorders that suppose an unacceptable risk according to investigators criteria.
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
* History of active primary immunodeficiency.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of AloCelyvir. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* Receipt of live attenuated vaccine within 30 days prior to the first dose of AloCelyvir. Note: Patients, if enrolled, should not receive live vaccine whilst receiving AloCelyvir and up to 30 days after the last dose of AloCelyvr.
* Female patients who are pregnant (confirmed with positive pregnancy test) or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose AloCelyvir.
* History of severe allergic reaction attributed to Celyvir or known hypersensitivity to any component of AloCelyvir dose composition.
* Resting ECG with clinically significant abnormal findings.
* Subjects with any one or more of the following:

  * History of myocardial infarction within 6 months prior to inclusion; patients with a history of myocardial infarction within 6 to 12 months prior to inclusion may be allowed following assessment
  * Unstable angina within 6 months prior to inclusion
  * Known significant cardiac disease (New York Heart Association [NYHA] classification of III or IV).
* History of stroke or transient ischemic attack within 6 months prior to inclusion.
* Evidence of any other disease, physical examination or laboratory finding giving reasonable suspicion of a disease or condition that puts the subject at high risk for treatment-related complication.
* Prior enrollment or treatment in a previous Alocelyvir clinical study regardless of treatment arm assignment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 6 months
  Objective Response Rate (ORR) is defined as the proportion of patients with at least one visit response of CR or PR that is confirmed at least 4 weeks later. Where PR is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters as long as criteria for PD are not met and CR is disappearance of all target lesions. Any pathological lymph nodes selected as target lesions must have a reduction in short axis to <10mm.
  Following RECIST 1.1 criteria, for non-randomised trials where response is the primary endpoint, confirmation of PR and CR is required to ensure responses identified are not the result of measurement error. ORR defined in this manner is a direct measure of drug antitumor activity, which can be evaluated in a single-arm study, providing an accurate assessment of a subrogate efficacy endpoint.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 3 months / 6 months
  Progression Free Survival (PFS) rate and Estimated PFS at 3, and 6-months according to RECIST 1.1 criteria For this protocol, PFS is defined as the time from enrollment until objective tumor progression or death according to section Primary Efficacy variable.Estimated PFS rate at 3 and 6-months are defined as the percentage of patients alive at 3 and 6-months from trial enrollment.
Overall Survival (OS) | 1 year / 2 years
  Overall Survival (OS) rate and Estimated Survival rate at 1, and 2-years. Overall Survival is defined as the time from enrollment until death from any cause. Estimated survival rate at 1 and 2 years are defined as the percentage of patients alive at 1st and 2nd year from trial enrollment.
Evaluate Safety | 2 years
  Evaluate Safety of the combination with AloCelyvir using NCI-CTCAE version 5.0. The safety objective of this trial is to characterize the safety and tolerability of AloCelyvir in subjects with mUM. The safety analysis will be based on subjects who experienced toxicities as defined by CTCAE, v5.0, the attribution to drug, time-of-onset, duration of the event, its resolution, and any concomitant medications administered will be recorded. AEs will be analysed including but not limited to all AEs, SAEs, fatal AEs, and laboratory changes. Furthermore, specific immunerelated adverse events (iris) will be collected and designated as immune related events of clinical interest (ECIs).

CONTACTS AND LOCATIONS:
Overall Officials: Josep M Piulats, MD, Phd, Principal Investigator — ICO, IDIBELL
Locations (1):
- ICO Hospitalet, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Osterlind A. Trends in incidence of ocular malignant melanoma in Denmark 1943-1982. Int J Cancer. 1987 Aug 15;40(2):161-4. doi: 10.1002/ijc.2910400206. PMID 3610385
- [Background] Jamison A, Bhatti LA, Sobti MM, Chadha V, Cauchi P, Kemp EG. Uveal melanoma-associated survival in Scotland. Eye (Lond). 2019 Nov;33(11):1699-1706. doi: 10.1038/s41433-019-0622-9. Epub 2019 Oct 25. PMID 31649344
- [Background] Bakalian S, Marshall JC, Logan P, Faingold D, Maloney S, Di Cesare S, Martins C, Fernandes BF, Burnier MN Jr. Molecular pathways mediating liver metastasis in patients with uveal melanoma. Clin Cancer Res. 2008 Feb 15;14(4):951-6. doi: 10.1158/1078-0432.CCR-06-2630. PMID 18281525
- [Background] Buder K, Gesierich A, Gelbrich G, Goebeler M. Systemic treatment of metastatic uveal melanoma: review of literature and future perspectives. Cancer Med. 2013 Oct;2(5):674-86. doi: 10.1002/cam4.133. Epub 2013 Sep 18. PMID 24403233
- [Background] Pons F, Plana M, Caminal JM, Pera J, Fernandes I, Perez J, Garcia-Del-Muro X, Marcoval J, Penin R, Fabra A, Piulats JM. Metastatic uveal melanoma: is there a role for conventional chemotherapy? - A single center study based on 58 patients. Melanoma Res. 2011 Jun;21(3):217-22. doi: 10.1097/CMR.0b013e3283457726. PMID 21467954
- [Background] Carvajal RD, Piperno-Neumann S, Kapiteijn E, Chapman PB, Frank S, Joshua AM, Piulats JM, Wolter P, Cocquyt V, Chmielowski B, Evans TRJ, Gastaud L, Linette G, Berking C, Schachter J, Rodrigues MJ, Shoushtari AN, Clemett D, Ghiorghiu D, Mariani G, Spratt S, Lovick S, Barker P, Kilgour E, Lai Z, Schwartz GK, Nathan P. Selumetinib in Combination With Dacarbazine in Patients With Metastatic Uveal Melanoma: A Phase III, Multicenter, Randomized Trial (SUMIT). J Clin Oncol. 2018 Apr 20;36(12):1232-1239. doi: 10.1200/JCO.2017.74.1090. Epub 2018 Mar 12. PMID 29528792
- [Background] Khoja L, Atenafu EG, Suciu S, Leyvraz S, Sato T, Marshall E, Keilholz U, Zimmer L, Patel SP, Piperno-Neumann S, Piulats J, Kivela TT, Pfoehler C, Bhatia S, Huppert P, Van Iersel LBJ, De Vries IJM, Penel N, Vogl T, Cheng T, Fiorentini G, Mouriaux F, Tarhini A, Patel PM, Carvajal R, Joshua AM. Meta-analysis in metastatic uveal melanoma to determine progression free and overall survival benchmarks: an international rare cancers initiative (IRCI) ocular melanoma study. Ann Oncol. 2019 Aug 1;30(8):1370-1380. doi: 10.1093/annonc/mdz176. PMID 31150059
- [Background] Robertson AG, Shih J, Yau C, Gibb EA, Oba J, Mungall KL, Hess JM, Uzunangelov V, Walter V, Danilova L, Lichtenberg TM, Kucherlapati M, Kimes PK, Tang M, Penson A, Babur O, Akbani R, Bristow CA, Hoadley KA, Iype L, Chang MT; TCGA Research Network; Cherniack AD, Benz C, Mills GB, Verhaak RGW, Griewank KG, Felau I, Zenklusen JC, Gershenwald JE, Schoenfield L, Lazar AJ, Abdel-Rahman MH, Roman-Roman S, Stern MH, Cebulla CM, Williams MD, Jager MJ, Coupland SE, Esmaeli B, Kandoth C, Woodman SE. Integrative Analysis Identifies Four Molecular and Clinical Subsets in Uveal Melanoma. Cancer Cell. 2017 Aug 14;32(2):204-220.e15. doi: 10.1016/j.ccell.2017.07.003. PMID 28810145
- [Background] Gezgin G, Dogrusoz M, van Essen TH, Kroes WGM, Luyten GPM, van der Velden PA, Walter V, Verdijk RM, van Hall T, van der Burg SH, Jager MJ. Genetic evolution of uveal melanoma guides the development of an inflammatory microenvironment. Cancer Immunol Immunother. 2017 Jul;66(7):903-912. doi: 10.1007/s00262-017-1991-1. Epub 2017 Apr 8. PMID 28391358
- [Background] van Essen TH, van Pelt SI, Bronkhorst IH, Versluis M, Nemati F, Laurent C, Luyten GP, van Hall T, van den Elsen PJ, van der Velden PA, Decaudin D, Jager MJ. Upregulation of HLA Expression in Primary Uveal Melanoma by Infiltrating Leukocytes. PLoS One. 2016 Oct 20;11(10):e0164292. doi: 10.1371/journal.pone.0164292. eCollection 2016. PMID 27764126
- [Background] Bronkhorst IH, Vu TH, Jordanova ES, Luyten GP, Burg SH, Jager MJ. Different subsets of tumor-infiltrating lymphocytes correlate with macrophage influx and monosomy 3 in uveal melanoma. Invest Ophthalmol Vis Sci. 2012 Aug 9;53(9):5370-8. doi: 10.1167/iovs.11-9280. PMID 22743317
- [Background] Qin Y, Petaccia de Macedo M, Reuben A, Forget MA, Haymaker C, Bernatchez C, Spencer CN, Gopalakrishnan V, Reddy S, Cooper ZA, Fulbright OJ, Ramachandran R, Wahl A, Flores E, Thorsen ST, Tavera RJ, Conrad C, Williams MD, Tetzlaff MT, Wang WL, Gombos DS, Esmaeli B, Amaria RN, Hwu P, Wargo JA, Lazar AJ, Patel SP. Parallel profiling of immune infiltrate subsets in uveal melanoma versus cutaneous melanoma unveils similarities and differences: A pilot study. Oncoimmunology. 2017 May 8;6(6):e1321187. doi: 10.1080/2162402X.2017.1321187. eCollection 2017. PMID 28680759
- [Background] Rothermel LD, Sabesan AC, Stephens DJ, Chandran SS, Paria BC, Srivastava AK, Somerville R, Wunderlich JR, Lee CC, Xi L, Pham TH, Raffeld M, Jailwala P, Kasoji M, Kammula US. Identification of an Immunogenic Subset of Metastatic Uveal Melanoma. Clin Cancer Res. 2016 May 1;22(9):2237-49. doi: 10.1158/1078-0432.CCR-15-2294. Epub 2015 Dec 28. PMID 26712692
- [Background] Alexander M, Mellor JD, McArthur G, Kee D. Ipilimumab in pretreated patients with unresectable or metastatic cutaneous, uveal and mucosal melanoma. Med J Aust. 2014 Jul 7;201(1):49-53. doi: 10.5694/mja13.10448. PMID 24999899
- [Background] Algazi AP, Tsai KK, Shoushtari AN, Munhoz RR, Eroglu Z, Piulats JM, Ott PA, Johnson DB, Hwang J, Daud AI, Sosman JA, Carvajal RD, Chmielowski B, Postow MA, Weber JS, Sullivan RJ. Clinical outcomes in metastatic uveal melanoma treated with PD-1 and PD-L1 antibodies. Cancer. 2016 Nov 15;122(21):3344-3353. doi: 10.1002/cncr.30258. Epub 2016 Aug 17. PMID 27533448
- [Background] Chandran SS, Somerville RPT, Yang JC, Sherry RM, Klebanoff CA, Goff SL, Wunderlich JR, Danforth DN, Zlott D, Paria BC, Sabesan AC, Srivastava AK, Xi L, Pham TH, Raffeld M, White DE, Toomey MA, Rosenberg SA, Kammula US. Treatment of metastatic uveal melanoma with adoptive transfer of tumour-infiltrating lymphocytes: a single-centre, two-stage, single-arm, phase 2 study. Lancet Oncol. 2017 Jun;18(6):792-802. doi: 10.1016/S1470-2045(17)30251-6. Epub 2017 Apr 7. PMID 28395880
- [Background] Dunn GP, Old LJ, Schreiber RD. The immunobiology of cancer immunosurveillance and immunoediting. Immunity. 2004 Aug;21(2):137-48. doi: 10.1016/j.immuni.2004.07.017. PMID 15308095
- [Background] Garcia-Castro J, Alemany R, Cascallo M, Martinez-Quintanilla J, Arriero Mdel M, Lassaletta A, Madero L, Ramirez M. Treatment of metastatic neuroblastoma with systemic oncolytic virotherapy delivered by autologous mesenchymal stem cells: an exploratory study. Cancer Gene Ther. 2010 Jul;17(7):476-83. doi: 10.1038/cgt.2010.4. Epub 2010 Feb 19. PMID 20168350
- [Background] Melen GJ, Franco-Luzon L, Ruano D, Gonzalez-Murillo A, Alfranca A, Casco F, Lassaletta A, Alonso M, Madero L, Alemany R, Garcia-Castro J, Ramirez M. Influence of carrier cells on the clinical outcome of children with neuroblastoma treated with high dose of oncolytic adenovirus delivered in mesenchymal stem cells. Cancer Lett. 2016 Feb 28;371(2):161-70. doi: 10.1016/j.canlet.2015.11.036. Epub 2015 Dec 3. PMID 26655276
- [Background] Cascallo M, Alonso MM, Rojas JJ, Perez-Gimenez A, Fueyo J, Alemany R. Systemic toxicity-efficacy profile of ICOVIR-5, a potent and selective oncolytic adenovirus based on the pRB pathway. Mol Ther. 2007 Sep;15(9):1607-15. doi: 10.1038/sj.mt.6300239. Epub 2007 Jun 19. PMID 17579575
- [Background] Suzuki K, Fueyo J, Krasnykh V, Reynolds PN, Curiel DT, Alemany R. A conditionally replicative adenovirus with enhanced infectivity shows improved oncolytic potency. Clin Cancer Res. 2001 Jan;7(1):120-6. PMID 11205899
- [Background] Garcia M, Moreno R, Gil-Martin M, Cascallo M, de Olza MO, Cuadra C, Piulats JM, Navarro V, Domenech M, Alemany R, Salazar R. A Phase 1 Trial of Oncolytic Adenovirus ICOVIR-5 Administered Intravenously to Cutaneous and Uveal Melanoma Patients. Hum Gene Ther. 2019 Mar;30(3):352-364. doi: 10.1089/hum.2018.107. Epub 2018 Nov 13. PMID 30234393
- [Background] Franco-Luzon L, Gonzalez-Murillo A, Alcantara-Sanchez C, Garcia-Garcia L, Tabasi M, Huertas AL, Chesler L, Ramirez M. Systemic oncolytic adenovirus delivered in mesenchymal carrier cells modulate tumor infiltrating immune cells and tumor microenvironment in mice with neuroblastoma. Oncotarget. 2020 Jan 28;11(4):347-361. doi: 10.18632/oncotarget.27401. eCollection 2020 Jan 28. PMID 32064039
- [Background] Rincon E, Cejalvo T, Kanojia D, Alfranca A, Rodriguez-Milla MA, Gil Hoyos RA, Han Y, Zhang L, Alemany R, Lesniak MS, Garcia-Castro J. Mesenchymal stem cell carriers enhance antitumor efficacy of oncolytic adenoviruses in an immunocompetent mouse model. Oncotarget. 2017 Jul 11;8(28):45415-45431. doi: 10.18632/oncotarget.17557. PMID 28525366
- [Background] Morales-Molina A, Gambera S, Cejalvo T, Moreno R, Rodriguez-Milla MA, Perise-Barrios AJ, Garcia-Castro J. Antitumor virotherapy using syngeneic or allogeneic mesenchymal stem cell carriers induces systemic immune response and intratumoral leukocyte infiltration in mice. Cancer Immunol Immunother. 2018 Oct;67(10):1589-1602. doi: 10.1007/s00262-018-2220-2. Epub 2018 Jul 31. PMID 30066102
- [Background] Cejalvo T, Perise-Barrios AJ, Del Portillo I, Laborda E, Rodriguez-Milla MA, Cubillo I, Vazquez F, Sardon D, Ramirez M, Alemany R, Del Castillo N, Garcia-Castro J. Remission of Spontaneous Canine Tumors after Systemic Cellular Viroimmunotherapy. Cancer Res. 2018 Sep 1;78(17):4891-4901. doi: 10.1158/0008-5472.CAN-17-3754. Epub 2018 Jul 10. PMID 29991502
- [Background] Kennedy S, Rice M, Toomey S, Horgan N, Hennessey BT, Larkin A. An insight into the molecular genetics of a uveal melanoma patient cohort. J Cancer Res Clin Oncol. 2018 Oct;144(10):1861-1868. doi: 10.1007/s00432-018-2705-6. Epub 2018 Jul 14. PMID 30008023
- [Background] Teng MW, Ngiow SF, Ribas A, Smyth MJ. Classifying Cancers Based on T-cell Infiltration and PD-L1. Cancer Res. 2015 Jun 1;75(11):2139-45. doi: 10.1158/0008-5472.CAN-15-0255. PMID 25977340
- [Background] Wolchok JD, Hoos A, O'Day S, Weber JS, Hamid O, Lebbe C, Maio M, Binder M, Bohnsack O, Nichol G, Humphrey R, Hodi FS. Guidelines for the evaluation of immune therapy activity in solid tumors: immune-related response criteria. Clin Cancer Res. 2009 Dec 1;15(23):7412-20. doi: 10.1158/1078-0432.CCR-09-1624. Epub 2009 Nov 24. PMID 19934295
- [Background] Nishino M, Giobbie-Hurder A, Gargano M, Suda M, Ramaiya NH, Hodi FS. Developing a common language for tumor response to immunotherapy: immune-related response criteria using unidimensional measurements. Clin Cancer Res. 2013 Jul 15;19(14):3936-43. doi: 10.1158/1078-0432.CCR-13-0895. Epub 2013 Jun 6. PMID 23743568
- [Background] Piulats JM, Espinosa E, de la Cruz Merino L, Varela M, Alonso Carrion L, Martin-Algarra S, Lopez Castro R, Curiel T, Rodriguez-Abreu D, Redrado M, Goma M, Rullan AJ, Calvo Gonzalez A, Berrocal-Jaime A. Nivolumab Plus Ipilimumab for Treatment-Naive Metastatic Uveal Melanoma: An Open-Label, Multicenter, Phase II Trial by the Spanish Multidisciplinary Melanoma Group (GEM-1402). J Clin Oncol. 2021 Feb 20;39(6):586-598. doi: 10.1200/JCO.20.00550. Epub 2021 Jan 8. PMID 33417511
- [Background] Piulats Rodriguez, J. M. et al. Phase II study evaluating ipilimumab as a single agent in the first-line treatment of adult patients (Pts) with metastatic uveal melanoma (MUM): The GEM-1 trial. J. Clin. Oncol. 32, 9033 (2014).
- [Background] Ruano D, Lopez-Martin JA, Moreno L, Lassaletta A, Bautista F, Andion M, Hernandez C, Gonzalez-Murillo A, Melen G, Alemany R, Madero L, Garcia-Castro J, Ramirez M. First-in-Human, First-in-Child Trial of Autologous MSCs Carrying the Oncolytic Virus Icovir-5 in Patients with Advanced Tumors. Mol Ther. 2020 Apr 8;28(4):1033-1042. doi: 10.1016/j.ymthe.2020.01.019. Epub 2020 Jan 21. PMID 32053771